CLINICAL TRIAL: NCT00560170
Title: Rho-kinase in Patients With Atherosclerosis: Effects of Statins A Randomized Clinical Trial Comparing Ezetimibe/Simvastatin and Simvastatin
Brief Title: Vascular Effects of Ezetimibe/Simvastatin and Simvastatin on Atherosclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: ASSISTANT PROFESSOR, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NCKUH-01/HR-95-112
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Atherosclerosis
Keywords: HMG-CoA Reductase Inhibitors; endothelial function; HMG-CoA Reductase Inhibitors on vascular protection
MeSH Terms: conditions — Atherosclerosis | interventions — Simvastatin; Ezetimibe; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- high dose statin (Experimental): 40mg of Simvastatin (n=20)
  Interventions: Drug: Simvastatin (Zocor)
- combination arm (Active Comparator): 10mg/10mg of Ezetimibe/Simvastatin (n=20)
  Interventions: Drug: 10mg/10mg of Ezetimibe/Simvastatin (Vytorin)

INTERVENTIONS:
Drug: Simvastatin (Zocor) — 40mg of Simvastatin (n=20) orally per-day for 28 days
  Other Names: Zocor
  Arms: high dose statin
Drug: 10mg/10mg of Ezetimibe/Simvastatin (Vytorin) — 10mg/10mg of Ezetimibe/Simvastatin (n=20) orally per-day for 28 days
  Other Names: Vytorin
  Arms: combination arm

SUMMARY:
Multiple clinical trials, using 3-hydroxy-3-methylglutaryl coenzyme A (HMG CoA) reductase inhibitors (statins), have shown benefit in the primary and secondary prevention of atherosclerotic complications. However, till now, there is an incomplete understanding of all the mechanisms of the biologic effects of statins beyond LDL cholesterol (LDL-C) reduction, but there is accumulating evidence that the Rho-GTP/Rho-Kinase pathway (Rho/Rho-K) plays an important role and may be a strategic therapeutic target in cardiovascular diseases. With similar LDL-C reduction ability, the availability of Ezetimibe offers the potential to begin to address the question whether some of the benefits conferred by statins may accrue independently of their effects on LDL-C lowering. A better understanding of the role of the Rho/Rho-kinase signaling pathway in the pathogenesis of atherosclerosis in human is essential. Inhibition of Rho/Rho-kinase by statins may explain some of the biological beneficial effects of statins observed in clinical trials. This study aims to translate into patients important experimental discoveries regarding the initiation of inflammation in atherosclerosis in an attempt to improve upon the present treatment of cardiovascular diseases.

DETAILED DESCRIPTION:
Study Design:

A single-blind controlled trial with two arms will be conducted at National Chen-Kung University Hospital (NCKUH). We will screen subjects with stable atherosclerosis to complete enrollment of 40 subjects in the study (see inclusion and exclusion criteria section below). A central pharmacist at NCKUH will randomize the patients to 40mg or Simvastatin (n=20) or 10mg/10mg of Ezetimibe/Simvastatin (n=20) for 28 days. If the patient is already on a statin a two-week washout period will be 2 weeks prior to trial initiation.

Primary Outcomes and measurement:

The primary outcomes are the mean changes in the Rho-kinase expression and activity in leukocytes in response to 40mg or Simvastatin (n=20) or 10mg/10mg of Ezetimibe/Simvastatin (n=20) over 28 days.

Secondary Outcomes and measurement:

The secondary outcomes are the correlation between the mean changes in Rho-kinase expression and activity in leukocytes and vascular tissue with the mean changes in LDL-C, hsCRP, and BAFMD, as well as its relation with clinical characteristics.

Subjects:

Participants will be recruited from the ambulatory clinics at the NCKUH Clinic.

Inclusion Criteria:

1. Male or female subjects aged 40 to 80 years
2. Documented stable atherosclerosis by angiography or vascular ultrasound (more that 20% luminal narrowing), peripheral arterial disease or type 2 diabetes mellitus (coronary heart disease (CHD) risk equivalent - Adult Treatment Program (ATP)-III guidelines)
3. LDL-cholesterol >100mg/dL (indication to treat with statin)
4. Written informed consent
5. Primary care physician authorization letter to participate in the study.

Exclusion criteria:

1. Inability to give consent
2. Pre-menopausal women
3. Current use of antibiotics, anti-inflammatory or immunosuppressant drugs
4. History of LFT >2 times the upper normal limit
5. History of myopathy / myositis or CPK > 10 times the upper normal limit
6. CPK above normal limits at study onset
7. Any evidence of inflammatory, infectious or neoplastic disease
8. History of CABG, PCI or acute ischemic syndrome in the preceding 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Male or female subjects aged 40 to 80 years
  2. Documented stable atherosclerosis by angiography or vascular ultrasound (more that 20% luminal narrowing), peripheral arterial disease or type 2 diabetes mellitus (coronary heart disease (CHD) risk equivalent - Adult Treatment Program (ATP)-III guidelines)
  3. LDL-cholesterol >100mg/dL (indication to treat with statin)
  4. Written informed consent
  5. Primary care physician authorization letter to participate in the study.
* Exclusion criteria:

  1. Inability to give consent
  2. Pre-menopausal women
  3. Current use of antibiotics, anti-inflammatory or immunosuppressant drugs
  4. History of LFT >2 times the upper normal limit
  5. History of myopathy / myositis or CPK > 10 times the upper normal limit
  6. CPK above normal limits at study onset
  7. Any evidence of inflammatory, infectious or neoplastic disease
  8. History of CABG, PCI or acute ischemic syndrome in the preceding 3 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
changes in the lipid profile change and Rho-kinase expression and activity | 28 days

SECONDARY OUTCOMES:
correlation between changes in Rho-kinase expression and activity with the changes in LDL-C, hsCRP and BAFMD | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Hong Chen, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Liu PY, Liu YW, Lin LJ, Chen JH, Liao JK. Evidence for statin pleiotropy in humans: differential effects of statins and ezetimibe on rho-associated coiled-coil containing protein kinase activity, endothelial function, and inflammation. Circulation. 2009 Jan 6;119(1):131-8. doi: 10.1161/CIRCULATIONAHA.108.813311. Epub 2008 Dec 15. PMID 19075102